CLINICAL TRIAL: NCT00110799
Title: A Double-Blind, Randomized, Placebo-Controlled, Multi-Centre, Dose-Ranging, Parallel Group, Phase II Study to Assess Efficacy, Safety/Tolerability, and Pharmacokinetics of a Thrombopoietin Receptor Agonist, SB-497115-GR, When Administered as 30, 50, and 75 mg Once Daily for 12 Weeks in Subjects With
Brief Title: SB497115 (Oral Thrombopoietin Receptor Agonist) Versus Placebo In Adults With Thrombocytopenia Due To Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPL102357
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Hepatitis C, Chronic; Hepatitis C; Thrombocytopenia
Keywords: thrombopoietin; platelets; Hepatitis C-related thrombocytopenia; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Thrombocytopenia; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Arm B (Active Comparator): SB-497115-GR 30mg administered orally daily for 12 weeks beginning 4 weeks prior to initiating 8 weeks of antiviral therapy and for 8 weeks during weekly antiviral therapy.
  Interventions: Drug: SB497115
- Arm C (Active Comparator): SB-497115-GR 50mg administered orally daily for 12 weeks beginning 4 weeks prior to initiating 8 weeks of antiviral therapy and for 8 weeks during weekly antiviral therapy.
  Interventions: Drug: SB497115
- Arm D (Active Comparator): SB-497115-GR 75mg administered orally daily for 12 weeks beginning 4 weeks prior to initiating 8 weeks of antiviral therapy and for 8 weeks during weekly antiviral therapy.
  Interventions: Drug: SB497115
- Arm A (Placebo Comparator): Placebo administered orally daily for 12 weeks beginning 4 weeks prior to initiating 8 weeks of antiviral therapy and for 8 weeks during weekly antiviral therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SB497115 — Approximately 160 subjects will be randomized equally to one of four treatment groups of approximately 40 subjects (A-D). Subjects will receive oral tablets of SB-497115-GR at 30mg, 50 mg, 75 mg or placebo administered once daily for a total of 12 weeks beginning 4 weeks prior to initiating 8 weeks of antiviral therapy and for 8 weeks during weekly antiviral therapy.
  Arms: Arm B; Arm C; Arm D
Other: Placebo — Placebo administered orally daily for 12 weeks beginning 4 weeks prior to initiating 8 weeks of antiviral therapy and for 8 weeks during weekly antiviral therapy.
  Arms: Arm A

SUMMARY:
SB497115 is an oral agent which activates the thrombopoietin receptor and increases platelet counts in healthy volunteers. This study is examining several different doses of SB497115 as a treatment for patients with chronic hepatitis C-related thrombocytopenia who are potential candidates for antiviral treatment with pegylated interferon and ribavirin. The study will be conducted in two phases, Parts 1 and 2. In Part 1, study subjects will be randomized to 4 weeks of SB-497115-GR or placebo administered daily without antiviral therapy. Subjects who successfully complete Part 1 (platelet count 70,000/µL for Pegasys and platelet count 100,000/µL for PEG-Intron) will then proceed to Part 2. In Part 2, subjects will receive an additional 8 weeks of SB-497115-GR or placebo administered daily with antiviral therapy.

DETAILED DESCRIPTION:
A Double-Blind, Randomized, Placebo-Controlled, Multi-Centre, Dose-Ranging, Parallel Group, Phase II Study to Assess Efficacy, Safety/Tolerability, and Pharmacokinetics of a Thrombopoietin Receptor Agonist, SB-497115-GR, when Administered as 30, 50, and 75 mg Once Daily for 12 weeks in Subjects with Chronic Hepatitis C-Related Thrombocytopenia who are Potential Candidates for Antiviral Treatment with Pegylated Interferon and Ribavirin.

ELIGIBILITY:
Inclusion criteria:

* Chronic low platelet count between 20,000 and <70,000/µL.
* Prior liver biopsy indicating chronic hepatitis within the previous 5 years or radiographic evidence of cirrhosis and / or endoscopic evidence of non-bleeding esophageal or gastric varices.

Exclusion criteria:

* History of heart attack or abnormal heart function.
* History of thrombosis within 1 year.
* History of alcohol or drug abuse or dependence within 1 year.
* Use of aspirin, aspirin-containing compounds, salicylates, antacids.
* History of HIV infection or active infection with Hepatitis B or C.
* Females who are pregnant.
* Patients using non-steroidal anti-inflammatory drugs during the study and within 3 weeks prior to starting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Treatment response, assessed by the proportion of subjects with a shift from baseline platelet count (20, 000 to <70,000µL) to =100,000/µL after 4 weeks of study treatment. | 4 weeks

SECONDARY OUTCOMES:
Mean increase in platelet counts and markers of thrombopoiesis. Safety and tolerability, population PK, pharmacodynamics. Effect of antiviral outcome measures during and after therapy. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (9):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Richmond, Virginia
- France (8):
  - GSK Investigational Site, Clermont Ferrand Cédex 1
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (6):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, San Juan, Puerto Rico
- United Kingdom (4):
  - GSK Investigational Site, Bristol, Gloucestershire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, London

REFERENCES:
- [Background] McHutchison JG, Dusheiko G, Shiffman ML, Rodriguez-Torres M, Sigal S, Bourliere M, Berg T, Gordon SC, Campbell FM, Theodore D, Blackman N, Jenkins J, Afdhal NH; TPL102357 Study Group. Eltrombopag for thrombocytopenia in patients with cirrhosis associated with hepatitis C. N Engl J Med. 2007 Nov 29;357(22):2227-36. doi: 10.1056/NEJMoa073255. PMID 18046027